CLINICAL TRIAL: NCT01445431
Title: A Randomized Controlled Trial on the Efficacy and Safety of Virgin Coconut Oil Compared to Mineral Oil in the Treatment of Uremic Xerosis
Brief Title: A Trial on the Efficacy and Safety of Virgin Coconut Oil Compared to Mineral Oil in the Treatment of Uremic Xerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Philippines (Other)
Responsible Party: Principal Investigator, Jacqueline Michelle G. de las Alas, M.D., Medical Officer III, University of the Philippines
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MED 2011-01-03-005
Record Dates: First submitted 2011-09-26; First posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Uremic Xerosis
MeSH Terms: interventions — Mineral Oil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virgin Coconut Oil (Experimental)
  Interventions: Other: Virgin Coconut Oil
- Mineral Oil (Active Comparator)
  Interventions: Other: Mineral Oil

INTERVENTIONS:
Other: Virgin Coconut Oil — Virgin coconut oil applied to the test site twice daily for four weeks
  Arms: Virgin Coconut Oil
Other: Mineral Oil — Mineral oil applied to the test site twice daily for four weeks
  Arms: Mineral Oil

SUMMARY:
Among adult patients with chronic kidney disease undergoing hemodialysis, what is the efficacy and safety of virgin coconut oil compared to mineral oil as a therapeutic moisturizer for uremic xerosis?

DETAILED DESCRIPTION:
Objectives of the Study: The general objective of this study is to assess the efficacy and safety of virgin coconut oil (VCO) compared to mineral oil as a therapeutic moisturizer for uremic xerosis. The specific objectives are as follows: 1) to determine and compare changes in the over-all dry skin score within and between treatment groups at baseline, 2 weeks-post and 4-weeks post application; 2) to quantitatively measure the following skin parameters at baseline, 2-weeks and 4-weeks post application (skin hydration using a corneometer, skin lipids using a sebumeter); 3) to determine and compare changes in quality of life scores within and between treatment groups at baseline, and 4-weeks post application; and 4) to identify the adverse effects of virgin coconut oil and mineral oil when used as moisturizer for uremic xerosis

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing maintenance hemodialysis who have mild to severe uremic xerosis

Exclusion Criteria:

* Patients with known hypersensitivity to the tests oils were excluded from the study as well as patients with open wounds, erosions, and ulcers on the test site and paraplegics and patients with altered sensation on the test sites.
* Patients with xerosis associated with other dermatologic conditions antedating renal failure were excluded from the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in baseline overall dry skin score | 4 weeks
Change in baseline corneometer readings | 4 weeks
  Measurement of skin hydration
Change in baseline sebumeter readings | 4 weeks
  Measurement of skin lipids

SECONDARY OUTCOMES:
Change in Quality of life scores | 4 weeks
Patient-assessed efficacy | 4 weeks
Adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Michelle G de las Alas, MD, Principal Investigator — University of the Philippines